CLINICAL TRIAL: NCT06083285
Title: Xinjiang Medical University of Affiliated Tumour Hospital
Brief Title: Impact of the CRRT Management Protocol on Prognostic Outcome in Patients With Septic Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiemuziya Maimaitirexiati, Associate Chief Physician, Xinjiang Medical University
Other Study IDs: XMaimaitirexiati
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: To Explore the Influence of CRRT Nursing Team Management Plan on the Prognosis of SAKI Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group
- Observation group
  Interventions: Other: Implement the CRRT specialist nursing group management program on the basis of routine care

INTERVENTIONS:
Other: Implement the CRRT specialist nursing group management program on the basis of routine care — Training the department nurses on CRRT related theoretical knowledge and operation skills; guiding the process of CRRT different treatment modes, solving CRRT nursing problems, evidence-based nursing guidance; consulting CRRT treatment and nursing related treatment, timely understanding the new progress; responsible for CRRT nursing quality control, etc.
  Groups: Observation group

SUMMARY:
The implementation of CRRT nursing team management program in the treatment of SAKI can significantly reduce the incidence of adverse events and complications in CRRT nursing, which has a positive role in improving the success rate of CRRT treatment and the clinical outcome of patients.

ELIGIBILITY:
Inclusion Criteria:

* The Guidelines for Emergency Treatment of Sepsis / Septic Shock in China (2018)[4]Diagnostic criteria for moderate sepsis; ② meets the Organization for Improving Global Kidney Disease Outcomes (KDIGO) Clinical Practice Guidelines: AKI[5]Relevant diagnostic criteria in; ③ received CRRT as indicated for CRRT; ④ in ICU for longer than 24 hours; ⑤ signed consent.

Exclusion Criteria:

* with chronic organ failure, or advanced malignancy; ② with previous history of chronic kidney disease, retrorenal urinary tract obstruction; ③ with incomplete clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 36 SAKI patients who were treated with CRRT in ICU of our hospital from February 2021 to August 2021 were set as the control group, and the routine bedside CRRT nursing management process was implemented in this stage; In addition, from September 2021 to March 2022, 40 SAKI patients who received CRRT treatment in our ICU were set as the observation group.The management plan of CRRT special nursing team was implemented to compare the incidence of non planned removal of CRRT, unplanned extubation and CRRT nursing related complications between the two groups, as well as the difference of coagulation function indexes before and 3 days after nursing.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
To explore the influence of CRRT nursing team management plan on the prognosis of SAKI patients. | 3-10 days
  The incidence of unplanned removal of CRRT, unplanned extubation and CRRT nursing related complications in the observation group were lower than those in the control group (P <0.05). Kaplan Meier survival curve showed that the survival rate of patients in the observation group was higher than that in the control group (P <0.05).

CONTACTS AND LOCATIONS:
Locations (1):
- Xinjiang Medical University of Affiliated tumour Hospital, Ürümqi, Xinjiang, China

IPD SHARING:
Plan to Share IPD: Undecided